CLINICAL TRIAL: NCT03402685
Title: Influence of Continuous Non-invasive Blood Pressure Measurement on Fetal Outcome After Caesarean Section ("ClearBirth")
Brief Title: Continuous Non-invasive Blood Pressure Measurement in C-section
Acronym: ClearBirth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Sascha Treskatsch, Deputy head of department Department of Anesthesiology and Operative Intensive Care Medicine, CCM and CVK; MD; PhD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ClearBirth
Record Dates: First submitted 2018-01-11; First posted 2018-01-18 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Cesarean Delivery Affecting Newborn; Cesarean Delivery Affecting Fetus; Cesarean Section Complications

STUDY DESIGN:
Intervention Model Description: Randomisation of patients using a randomisation list drawn up by an independent statistician in either NIBP or ClearSight group. In both groups, the above-mentioned standard procedure according to SOP and also the non-invasive continuous blood pressure measurement to improve blood pressure monitoring with the ClearSight system, so that all patients are monitored by both monitoring systems. In the NIBP Group, anaesthetists are blinded against the ClearSight measurement. In the ClearSight group, anaesthetists are blinded against the NIBP measurement. Blinding is achieved by completely covering the measured values of the other method.
Who Masked: Participant, Outcomes Assessor
Masking Description: The statistician is not informed about the group names, the APGAR scores are awarded by independent neonatologists/pediatricians and gynaecologists.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NIBP-Group (No Intervention): NIBP will be shown, ClearSight will be covered.
- ClearSight-Group (Experimental): ClearSight will be shown, NIBP will be covered.
  Interventions: Device: ClearSight

INTERVENTIONS:
Device: ClearSight — Patients in the intervention group receive management of volume and vasopressor settings according to the non-invasive ClearSight system.
  Other Names: non-invasive continous blood pressure measurement
  Arms: ClearSight-Group

SUMMARY:
The caesarean section is a frequently performed procedure in obstetrics and accounts for about 30% of all births in Germany. 55% to 68% of all caesarean sections are performed under spinal anesthesia. A possible side effect of spinal anesthesia is arterial hypotension with a prevalence of 70% to 80%. A placental hypoperfusion in the context of a reduced preload due to hypotension can reduce the fetal outcome. Early diagnosis and treatment of the hypotensive episode could reduce and at best prevent increased fetal morbidity.

Due to their invasiveness due to the necessity of puncturing a distal artery of the extremity and the insertion of a catheter, established continuous blood pressure measurement procedures have disadvantages such as potential circulatory disorders of the hand, infections, bleeding and thrombosis and are therefore often not indicated in the context of an elective sectio. Non-invasive procedures such as NIBP, however, are discontinuous and may make a timely diagnosis of hypotension more difficult and delay therapy. The ClearSightTM system, which allows a continuous non-invasive blood pressure measurement, has been used in hip and knee joint surgery. There, a good correlation with invasive blood pressure measurements was found, particularly with regard to systolic and mean arterial pressure. An application in obstetrics has not yet been investigated. Due to the continuous measurement provided by ClearSightTM, continuous monitoring of blood pressure appears to be ensured, so that a faster reaction to previously undetected fluctuations in blood pressure can be expected compared to interval measurement.

DETAILED DESCRIPTION:
The determination of arterial blood pressure is a basic monitoring measure during spinal anaesthesia in obstetrics for the operative delivery of the child via the caesarean section. Adequate arterial blood pressure is essential to ensure adequate placental perfusion, sufficient cerebral perfusion pressure of the mother and is the basis for any hemodynamic optimization to significantly improve patient outcome.

Up to now, two standard methods for determining blood pressure have always been the oscillating non-invasive, intermittent blood pressure measurement (NIBP) and the invasive continuous blood pressure measurement (IBP). The NIBP derives blood pressure values using upper arm cuffs at defined intervals. As a result, no continuous measurement is possible and nerve damage and pain are risks of this method. The indication for the establishment of IBP is often not given due to potential side effects such as aneurysm formation, infections, thrombosis and circulatory impairment of the hand. The application of a novel non-invasive, patch-clamp-based continuous blood pressure measurement system (ClearSightTM, Edwards Lifesciences Corporation, Irvine, California, USA) promises to combine the advantages of NIBP, namely non-invasiveness and IBP, the continuous pressure measurement. So far, there have been no randomized, controlled trials for application. Spinal anesthesia is a widespread anaesthetic procedure for performing Caesarean sections. Within the clinical standard, an intermittent blood pressure measurement is used at intervals of 2 to 5 minutes. Continuous invasive blood pressure measurement is not a standard procedure.

Standard procedure: The standard procedure corresponds to the SOPs of the Clinic for Anaesthesiology and intensive care medicine. After admission to the operating room, the patient is monitored by means of a 3-channel ECG and pulse oximetry. The NIBP measurement by means of an upper arm cuff is carried out intermittently with a measurement interval of 2 minutes according to SOP (standard operating procedure) and is continued until the umbilical cord of the fetus is removed. Subsequently, a peripheral venous access is applied and 500 ml of full electrolyte solution are infused. Subsequently, the spinal anesthesia is applied in a seated position. Size-adapted 1.6 - 2.0 ml hyperbaric bupivacaine 0.5%, 0.1 mg morphine and 5 µg sufentanil are used. According to SOP, local skin infiltration with lidocaine 1% is carried out. After application of the spinal anaesthesia, the patient is positioned in a supine position with the operating table tilted 15° to the left. If the systolic blood pressure drops below 100 mmHg or by more than 20 % of the initial value, 100 µg phenylephrine is applied. After a sufficient entry into action (target height according to SOP TH4) the Caesarean section is performed. After birth, APGAR values are recorded after 1,5 and 10 minutes, and umbilical cord blood gas analysis is performed.

Study procedure: Randomisation of patients based on a randomisation list drawn up by an independent statistician in either NIBP or ClearSight group. In both groups, the above-mentioned standard procedure according to SOP and also the non-invasive continuous blood pressure measurement to improve blood pressure monitoring with the ClearSight? system, so that all patients are monitored by both monitoring systems. In the NIBP Group, anaesthetists are blinded against the ClearSight measurement. In the ClearSight group, anaesthetists are blinded against the NIBP measurement. Blinding is achieved by completely covering the measured values of the other method. (please describe in detail). The installation of the measuring sensors does not involve any risks for patients.

ELIGIBILITY:
Inclusion Criteria:

* Female patients who receive a caesarean section under spinal anaesthesia
* Presence of the written declaration of consent
* Age >/= 18 years
* No participation in another prospective intervention study during participation in this study

Exclusion Criteria:

* Symptomatic heart failure NYHA >/= III (New York Heart Association)
* Symptomatic valve disease (stenosis/insufficiency) >/= II°
* Liver failure CHILD >/= B
* Acute or chronic renal impairment requiring dialysis
* (pre-)clampsia
* HELLP syndrome
* current or previous alcohol or drug abuse
* Psychiatric diseases
* sepsis
* side difference of the blood pressure measured during screening for vascular pathologies with blood pressure >12mmHg by means of NIBP

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Time | duration of surgery (an average of 2 hours)
  Mean difference in time to detection and treatment of hypotension between continuous non-invasive (ClearSight) blood pressure measurement and NIBP, determined by the area under the curve (AUC) of latency between hypotension and therapy.

SECONDARY OUTCOMES:
APGAR-1 | after delivery (an average of 1 minute)
  APGAR value 1 minute after delivery
APGAR-5 | after delivery (an average of 5 minutes)
  APGAR value 5 minutes after delivery
APGAR-10 | after delivery (an average of 10 minutes)
  APGAR value 10 minutes after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Sascha Treskatsch, MD, Prof, Principal Investigator — Charite
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No